CLINICAL TRIAL: NCT01798420
Title: The Impact of Corticosteroid Treatment on Hemoglobin A1C Levels in Diabetic Patients With COPD Exacerbation
Brief Title: Corticosteroids and Hemoglobin A1C Levels in Diabetic Patients With COPD Exacerbation
Status: Completed | Type: Observational
Sponsor: The Nazareth Hospital, Israel (Other)
Responsible Party: Principal Investigator, George Habib, Head, Rheumatology clinic, Nzareth hospital, Nzareth, The Nazareth Hospital, Israel
Other Study IDs: Hb-A1C-2012
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes; Chronic Obstructive Pulmonary Disease
Keywords: COPD; Diabetes; steroids; Hemoglobin A1C DIFFERENCE
MeSH Terms: conditions — Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Corticosteroid
- non-corticosteroid group

SUMMARY:
Corticosteroid treatment in diabetic patients admitted for COPD exacerbation are expected to significantly increase hemoglobin A1C levels

DETAILED DESCRIPTION:
HbA1C levels were evaluated in diabetic patients with COPD exacerbation on admission to the hospital and 3-months later. Demographic, clinical, laboratory variables and total steroid dose were documented. Age- and sex-matched group of diabetic patients with COPD who were admitted for other reasons, were asked to participate as a control group. Mann-Whitney and Chi square/Fischer's exact tests were used to compare between the parameters of the two groups. Wilcoxon signed rank test was used to compare between HbA1C levels at baseline and 3 months later. Multi-variate linear regression analysis was used to find predictors for increase in HbA1C levels in the patients' group.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with COPD exacerbation

Exclusion Criteria:

* Patients treated with steroids during the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with COPD ecaxerbation who are admitted to the hospital
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C LEVEL | 3 MONTHS

SECONDARY OUTCOMES:
Glucose levels | 3 months

OTHER OUTCOMES:
Weight | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of medicine, Nzareth, Nazareth, Israel